CLINICAL TRIAL: NCT04010123
Title: Post-Market Clinical Follow Up of Rotarex®S Catheter
Status: Completed | Type: Observational
Sponsor: Straub Medical AG (Industry)
Responsible Party: Sponsor
Other Study IDs: PMCF-001
Record Dates: First submitted 2019-05-10; First posted 2019-07-08 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2020-12

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Atherectomy; Thrombectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Atherectomy/Thrombectomy — Percutaneous transluminal removal of thrombotic, thromboembolic and atherothrombotic material from fresh, subacute and chronic occlusions of blood vessels in native blood vessels or vessels fitted with stents, stent grafts or native or artificial bypasses.

SUMMARY:
Post-Market Clinical Follow Up of the Rotarex®S Catheter

DETAILED DESCRIPTION:
A prospective, multi-center, non-randomized, multiple cohorts, observational, post market clinical follow-up study of the Rotarex®S Catheter to evaluate the safety, technical performance and medical efficacy of the Rotarex®S Catheter as a stand-alone and adjunctive therapy for the treatment of acute, subacute and chronic occlusions and sub-occlusions of arteries outside the cardiopulmonary, coronary and cerebral circulations, in accordance with Rotarex®S Catheter intended use.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is ≥18 years old at the time of consent.
2. Subject has provided written informed consent prior to participation in the study, understands the purpose of this study and agrees to comply with all protocol-specified examinations and follow-up appointments.
3. Female patients of childbearing potential have negative pregnancy test ≤7 days before the procedure.
4. Documented symptomatic peripheral arterial disease.
5. Acute, subacute and chronic (sub-) occlusion, with ≥ 90% stenosis in native arteries and/or stents / stent grafts and/or Bypass grafts and/or AV Fistula (Dialysis access).
6. De novo or re-occluded lesion.
7. Vessel and/or stent diameter within treatable range as per Instruction For Use.
8. Occlusion crossed intraluminally by a guidewire.

   For patients requiring lower limb intervention:
9. Patient presenting with a category from 2 to 5 according to the Rutherford classification for chronic limb ischemia or a category from I to IIb according to the Rutherford classification for acute limb ischemia.

Exclusion Criteria:

1. Life expectancy < 2 years.
2. Pregnant or nursing a child.
3. Contraindication, intolerance, or allergy to contrast media that, in the opinion of the investigator, cannot be adequately pre-medicated.
4. Myocardial infarction within 60 days prior to index procedure.
5. History of severe trauma and/or sepsis within 60 days prior to index procedure.
6. Cerebrovascular accident (CVA) or Transient Ischemic Attack (TIA) within 60 days prior to index procedure.
7. Evidence of intracranial or gastrointestinal bleeding or intracranial aneurysm within 90 days prior to index procedure.
8. Abnormal electrocardiogram or blood test results and/or any other factor that would increase risk by participating in the study in the opinion of the investigator.
9. Target lesion not crossed with guidewire or extraluminal guidewire crossing (even if in short segments only).
10. Additional lesion that is located >3cm away from the target lesion
11. Treatment plan of the target lesion includes laser, brachytherapy, or atherectomy other than the Rotarex®S Catheter.
12. Patient is currently participating in another investigational drug or device study that has not reached the primary endpoint.
13. Patients contraindicated for antiplatelet therapy, anticoagulants or thrombolytics.
14. Patients with uncorrected bleeding disorders.
15. Thrombophlebitis or deep vein thrombosis within the past 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute / Subacute / Chronic occlusions (Thrombotic / Thromboembolic / Atherothrombotic) of Native Arteries, Stents and Stents-grafts, Bypass grafts and AV-Fistula (Dialysis access))
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2019-07-17 (Actual); Primary Completion 2022-10-26 (Actual); Study Completion 2022-10-26 (Actual)

PRIMARY OUTCOMES:
Freedom from major adverse events (MAE) | 30 days
  Defined as clinically driven target lesion revascularization (TLR), any death and any unplanned major amputation of the index limb.

SECONDARY OUTCOMES:
(MAE) Major adverse events Rate | 6, 12 and 24 months
  Defined as clinically driven target lesion revascularization (TLR), any death and any unplanned major amputation of the index limb.
Technical success | Day 1
  defined as the ability to cross and treat the target lesion with the Rotarex®S Catheter to achieve residual angiographic stenosis no greater than 50% directly after Rotarex®S Catheter use.
Freedom of Target Lesion Revascularization (TLR) | 12 Months
  Freedom of Target Lesion Revascularization (TLR)
Freedom of Target Vessel Revascularization (TVR) | 1, 6, 12 and 24 Months
  Freedom of Target Vessel Revascularization (TVR)
Incidence of clinically significant Rotarex®S Catheter -related distal embolization requiring further treatment with pharmacologic or mechanical devices (except treating with intravascular nipride or nitroglycerin). | From start to end of procedure
  Rotarex®S Catheter -related distal embolization requiring further treatment with pharmacologic or mechanical devices (except treating with intravascular nipride or nitroglycerin).
Incidence of Rotarex®S Catheter -related perforations. | From start to end of procedure
  Rotarex®S Catheter -related perforations.
Clinical success | 1, 6, 12 and 24 months
  Defined as clinical category improvement in the Rutherford Class at 1, 6, 12 and 24 months with reference to the baseline value.
Hemodynamic success | 30 days
  Defined as a > 0.15 improvement in ABI (ankle-brachial index) at 30 days with reference to the baseline value.
Primary patency at 1, 6, 12 and 24 months. | 1, 6, 12 and 24 months
  Defined as freedom from >50% restenosis as indicated by an independently verified duplex ultrasound peak systolic velocity ratio (PSVR) < 2.5 in the target vessel with no clinically driven target lesion revascularization (TLR).
Walking improvement at 1, 6, 12 and 24 months assessed by Vascu Quality of Life Questionnaire (VQ-6). | 1, 6, 12 and 24 months
  Walking improvement assessed by Vascu Quality of Life Questionnaire (VQ-6)
Quality of Life improvement at 1, 6, 12 and 24 months assessed by Questionnaire. (EQ5D-3L) | 1, 6, 12 and 24 months
  Improvement of quality of life assessed by Questionnaire (EQ5D-3L)
Duration of hospital stay for index procedure [days]. | Duration of hospital stay, up to 12 weeks
  Number of day from admission to discharge from hospital.
Duration of ICU stay for index procedure [days]. | Duration of ICU stay, up to 12 weeks
  Number of day from admission to discharge from intensive care unit.
Procedural success | From start to end of procedure
  Successful revascularization of target lesion defined as ≤30% residual angiographic diameter stenosis following Rotarex®S Catheter treatment ± adjunctive treatment.
Successful use of Arterio Venous-Fistula as dialysis access, defined as successful use of the fistula for dialysis on at least one occasion. | Up to 14 days
  Only for patient subject to Arterio Venous-Fistula treatment with Rotarex®S Catheter.
Number of patients whose hemodialysis is efficient at 1, 6, 12 and 24 months without needing further treatment of the stenotic site after Rotarex®S treatment of the Arterio Venous-Fistula. | 1, 6, 12 and 24 months
  Only for patient subject to Arterio Venous-Fistula treatment with Rotarex®S Catheter.
(SAEs) Serious Adverse events Rate | 6, 12 and 24 months
  SAEs as defined per ISO 14155.
Procedure-related Adverse events Rate | 6, 12 and 24 months
  Procedure-related AEs as defined per ISO 14155.
(ADEs) Adverse device effects Rate | 6, 12 and 24 months
  Adverse device effects (ADEs) as defined per ISO 14155.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lichtenberg, Dr. med., Study Director — Klinikum Hochsauerland GmbH
Locations (13):
- Angiocentrum Příbram, Příbram, Czechia
- East-Tallinn Central Hospital, Tallinn, Estonia
- CHU - Hôpital François-Mitterrand, Dijon, France
- Germany (9):
  - Klinikum Hochsauerland GmbH, Arnsberg
  - Universitäts-Herzzentrum Freiburg - Bad Krozingen, Bad Krozingen
  - Klinikum Friedrichshafen, Friedrichshafen
  - Universitätsklinik Leipzig, Leipzig
  - Bonifatius Hospital, Lingen
  - Universitätsklinikum Münster, Münster
  - Elblandklinikum Radebeul, Radebeul
  - Elblandklinikum Riesa, Riesa
  - Kreiskrankenhaus Torgau "Johann Kentmann", Torgau
- Ospedale P. Pederzoli - Casa di Cura Privata Spa, Peschiera del Garda, Italy